CLINICAL TRIAL: NCT03868696
Title: Ultrasound Directed Reduction of Colles Type Distal Radial Fractures in ED (UDiReCT)
Acronym: UDiReCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: Royal College of Emergency Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 251149
Record Dates: First submitted 2019-02-20; First posted 2019-03-11 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-03

CONDITIONS: Radius Distal Fracture; Colles' Fracture
Keywords: Ultrasound; Manipulation under anaesthesia; Emergency Department
MeSH Terms: conditions — Wrist Fractures; Colles' Fracture; Emergencies

STUDY DESIGN:
Intervention Model Description: 1:1 randomised stratified by centre
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Sham ultrasound will be conducted in control group with screen off and facing away from participant.
  Active US screen will also be turned away from participant in the US allocated group and no discussion allowed about the image.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MUA with sham ultrasound (Sham Comparator): Participants will undergo standard manipulation (MUA) of wrist fracture with sham ultrasound (screen concealed from participants)
  Interventions: Procedure: MUA with sham ultrasound
- MUA with active ultrasound (Experimental): Participants will undergo standard manipulation (MUA) of wrist fracture with active ultrasound (screen concealed from participants)
  Interventions: Procedure: MUA with active ultrasound

INTERVENTIONS:
Procedure: MUA with sham ultrasound — Standard MUA with sham ultrasound
  Arms: MUA with sham ultrasound
Procedure: MUA with active ultrasound — Standard MUA guided by ultrasound
  Arms: MUA with active ultrasound

SUMMARY:
This is a limited two centre randomized controlled feasibility trial towards a larger definitive trial designed to assess whether bed side ultrasound can reduce the rate of surgical fixation following emergency department manipulation of Colles' type wrist fractures. UDiReCT will mirror the proposed design of the definitive trial but will report feasibility data such as recruitment rate, data completeness and reliability of potential definitive trial outcome measures.

DETAILED DESCRIPTION:
Wrist fractures are one of the most common fractures encountered in the Emergency Department (ED). These injuries most frequently happen in people who have fallen onto an outstretched hand and can result in deformity ('displacement') of the broken bone. These 'displaced' (Colles' types of distal radial) fractures can result in long term deformity and problems using the wrist. To prevent this, patients with displaced fractures often undergo manipulation of their fractures, to straighten the wrist, using local anaesthetic or sedation techniques in ED before a plaster cast is applied.

Unfortunately, if ED fracture manipulation is inadequate or the position later 'slips', which can occur in the first 1-2 weeks even in cast, then the patient will need to be admitted to hospital for surgical fixation. Local audit data suggests this affects up to a third of these patients and is a significant additional social and economic burden for patients and healthcare services.

Reducing these fractures as precisely as possible might reduce the subsequent need for surgery. However, ED fracture manipulations are typically done 'blind' with check x-rays after casting, making re-manipulation time consuming with prolonged local anaesthetic times or need for re-sedation. Portable, bedside ultrasound is available in most departments and has been used to guide fracture reduction but it is not known how effective this is nor is it in routine use. Providing this evidence would require a large, multi-centre randomized controlled trial (RCT) trial.

This project aims to determine whether such a trial comparing current practice with ultrasound guided reductions is justified and feasible. This will be done by running a feasibility RCT across two United Kingdom (UK) hospital sites to assess recruitment rates and trial procedures. The investigators hope to recruit about 60 patients in 6 months. This trial will include adults' aged 18 years and older, with Colles' type of distal radial fractures requiring manipulation in ED.

ELIGIBILITY:
Inclusion Criteria:

* Adults with Colles' type fractures of the distal radius undergoing fracture manipulation in the ED
* UDiReCT Trial trained staff available

Exclusion Criteria:

* Age under 18
* Volar displaced (Smith's) type fractures (well established as being unstable and requiring surgical treatment)
* Unable or unwilling to give informed consent
* Unable or unwilling to be followed up (e.g. orthopaedic follow up in another region)
* Major trauma with other injuries and ISS (Injury Severity Score) >16
* Urgent manipulation required due to neurovascular or skin compromise
* Open fractures or those with associated nerve or tendon involvement (affect functional outcome)
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Participant recruitment rate | 6 months
  Number of participants recruited over the duration of the study

SECONDARY OUTCOMES:
Data completeness. | 6 months
  The reliability and completeness of data proposed to be collected in a future definitive trial. Measured by the proportion of database fields completed by the end of the study

OTHER OUTCOMES:
Emergency Department (ED) manipulation under anaesthesia (MUA) failure rate | 6 months
  The proportion (%) of cases having undergone surgical fixation of the index fracture after ED MUA, within 6 weeks of injury . This is the proposed outcome for a definitive trial.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Emergency Department, Exeter, Devon
  - Barking, Havering and Redbridge University Hospitals Nhs Trust, London

REFERENCES:
- [Derived] Malik H, Wood D, Stone O, Gough A, Taylor G, Knapp KM, Heggs D, Appelboam A. Ultrasound Directed Reduction of Colles' type distal radial fractures in ED (UDiReCT): a feasibility randomised controlled trial. Emerg Med J. 2023 Nov 28;40(12):832-839. doi: 10.1136/emermed-2023-213279. PMID 37890981